CLINICAL TRIAL: NCT02534116
Title: A Comparison of Incisional Negative-Pressure Wound Therapy Versus Conventional Dressings Following Abdominal Surgery: A Randomized-Controlled Trial
Brief Title: A Comparison of Incisional Negative-Pressure Wound Therapy Versus Conventional Dressings Following Abdominal Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never began
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1511016790
Record Dates: First submitted 2015-08-13; First posted 2015-08-27 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Abdominal Reconstruction
Keywords: abdominal reconstruction
MeSH Terms: interventions — Negative-Pressure Wound Therapy; Therapeutics; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vacuum-assisted closure (VAC) therapy (Experimental): Following closure of the incision, patients will have incisional vacuum-assisted closure (VAC) therapy performed.
  Interventions: Procedure: Vacuum-assisted closure (VAC) therapy
- Gauze dressing (Active Comparator): Following closure of the incision, patients will either have a gauze dressing placed over the incision.
  Interventions: Procedure: Gauze dressing

INTERVENTIONS:
Procedure: Vacuum-assisted closure (VAC) therapy — Following closure of the incision, patients will either have a gauze dressing placed over the incision (control group), or incisional vacuum-assisted closure (VAC) therapy. The dressing will be removed over a time period of 2 to 5 days after surgery. The gauze dressing will be removed at 2 days and the wound VAC will be removed at 5 days.
  Other Names: Negative-pressure wound therapy (NPWT)
  Arms: Vacuum-assisted closure (VAC) therapy
Procedure: Gauze dressing — Following closure of the incision, patients will either have a gauze dressing placed over the incision (control group), or incisional vacuum-assisted closure (VAC) therapy. The dressing will be removed over a time period of 2 to 5 days after surgery. The gauze dressing will be removed at 2 days and the wound VAC will be removed at 5 days.
  Other Names: standard care
  Arms: Gauze dressing

SUMMARY:
The purpose of this study is to compare outcomes between incisional negative-pressure wound vacuum-assisted closure (VAC) therapy versus conventional dressings following abdominal surgery.

DETAILED DESCRIPTION:
This study will prospectively compare rates of wound complications using incisional negative pressure wound therapy versus conventional dressings following abdominal reconstruction.

Patients will undergo abdominal surgery (panniculectomy, abdominoplasty, ventral hernia repair, or autologous flap reconstruction using abdominal donor tissue). Following closure of the incision, patients will either have a gauze dressing placed over the incision (control group), or incisional vacuum-assisted closure (VAC) therapy. The dressing will be removed over a time period of 2 to 5 days after surgery. The gauze dressing will be removed at 2 days and the wound VAC will be removed at 5 days. After this time, the wound will be assessed for signs of infection, seroma, hematoma, skin and fat necrosis, skin dehiscence, and hernia during the follow-up appointments.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in this study are patients undergoing abdominal reconstruction, which includes panniculectomy, abdominoplasty, ventral hernia repair and patients undergoing autologous flap reconstruction using abdominal donor tissue.

Exclusion Criteria:

* Patients will be excluded from study if they have an actively infected wound involving the incision, abdominal malignancy, a history of enteric fistula formation, or a bleeding disorder.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12 (Estimated); Primary Completion 2016-10 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Post Operative Wound Complications | Between 2 and 5 days following surgery
  Post-operative wound complications (infection, seroma, hematoma, skin and fat necrosis, skin dehiscence, and hernia) will be assessed at 2 days for gauze patients and at 5 days for VAC patients. This outcome will be assessed based on the clinical examination by the surgeon following removal of the wound dressing. There is no defined assessment tool for this outcome as clinical observation is the standard in these procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Persing, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, Section of Plastic Surgery, New Haven, Connecticut, United States